CLINICAL TRIAL: NCT01418092
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled, 12-week Study to Evaluate the Safety and Efficacy of ALKS 37 in Subjects With Opioid-induced Constipation
Brief Title: ALK37-007: Evaluation of Safety and Efficacy of ALKS 37 (RDC-1036) in Adults With Opioid-induced Constipation (OIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK37-007
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: OIC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Capsules for oral administration
  Interventions: Drug: Placebo
- ALKS 37 (Experimental): Capsules for oral administration
  Interventions: Drug: ALKS 37

INTERVENTIONS:
Drug: ALKS 37 — Capsules for oral administration
  Arms: ALKS 37
Drug: Placebo — Capsules for oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ALKS 37 when administered daily to adults with OIC.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age at time of consent
* Have a body mass index (BMI)of 19 to 35 kg/m2 at screening
* Are receiving prescribed opioid medication for the management of chronic, non-cancer pain
* Meet the criteria of OIC
* Agree to use an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Pregnancy and/or currently breastfeeding
* Clinically significant medical condition or illness (other than the condition for which the pain medication is being prescribed)
* Receiving treatment with opioid therapy for cancer-related pain, abdominal pain, scleroderma, and/or for the management of drug addiction
* Any gastrointestinal (GI) disorder (other than opioid-induced constipation) or GI structural abnormality known to affect bowel transit, produce GI obstruction, or contribute to bowel dysfunction
* Use of naloxone, Subutex or Suboxone, Revia, Vivitrol, Relistor, or Entereg starting 15 days before the first study visit following screening until the end of the study
* Participation in a clinical trial of a pharmacological agent within 30 days before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly average of complete spontaneous bowel movements during treatment | Weeks 1 through 4 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh-Pemberton, M.D., Study Director — Alkermes, Inc.
Locations (13):
- United States (13):
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Daytona Beach, Florida
  - Alkermes Investigational Site, Plantation, Florida
  - Alkermes Investigational Site, Marietta, Georgia
  - Alkermes Investigational Site, Indianapolis, Indiana
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Willingboro, New Jersey
  - Alkermes Investigational Site, Raleigh, North Carolina
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Bellevue, Washington